CLINICAL TRIAL: NCT03897634
Title: Clinical Trial of Roger Adaptive Digital Technology
Brief Title: Remote Microphone Candidacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Phonak AG, Switzerland (Industry)
Responsible Party: Principal Investigator, Pamela Souza, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0053453
Record Dates: First submitted 2019-03-20; First posted 2019-04-01 (Actual); Results first posted 2021-05-28 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Assistive Listening Device (ALD); Hearing in Noise
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: Within-subject design: Baseline assessments compared to post-trial results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experiences Hearing Aid user (Experimental): Single arm study, all participants in this arm. Participants will be experienced hearing aid users.
  Interventions: Device: Remote Microphone

INTERVENTIONS:
Device: Remote Microphone — Experienced hearing aid users will be trained on and use a remote microphone for 30 days. Pre- and Post- measures will be taken to determine benefit. Participant characteristics will also be assessed (such as self-efficacy) to explore personality factors that may contribute to benefit from devices.
  Other Names: Roger Select

SUMMARY:
Despite improvements in digital hearing aid technology, many hearing aid users continue to report difficulty understanding speech in challenging listening environments. Remote microphones have been shown to provide benefit in the most common of these challenging listening environments: distant speakers, background noise, and reverberation. Despite demonstrated benefit, there is a low rate of remote microphone use among adult hearing aid users. One reason for low uptake may be an uncertainty among hearing healthcare providers and potential users regarding expected clinically relevant benefit. This clinical trial will attempt the following:

1. To describe the range of remote microphone benefit among adults with mild-to-moderate sensorineural hearing loss
2. To determine specific individual factors beyond the audiogram that are associated with greater benefit from remote microphones

DETAILED DESCRIPTION:
2.0 Background / Literature Review / Rationale for the study:

Even when wearing well-fit hearing aids, many individuals with hearing loss continue to report difficulty communicating in background noise is one of the most common complaints of individuals with hearing loss. Directional microphones can improve speech perception in noise, but often fail to provide benefit in cases where the talker is distant from the listener, where there are multiple or moving noise sources, or in reverberation. Digital noise reduction may reduce listening effort and improve listening comfort, but has minimal effect on speech perception.

Placing the microphone in close proximity to the talker reduces the effective distance between speaker and listener, compensating for the effects of background noise and reverberation on the target signal. Use of a remote microphone can significantly improve signal-to-noise ratio (SNR), thereby improving speech perception in noise and at a distance. Recent studies demonstrated that remote-microphone devices that utilize adaptive digital technology (i.e, Roger) provide significantly more benefit for speech understanding in noise than non-adaptive remote microphones. Those advantages are likely related to the adaptive nature of the device, whereby the microphone gain varies according to the level of noise in the environment. In addition, interference is reduced via transmission of short digital bursts (160 μs) across a range of channels (2.4-2.4835 GHz). Further, the ability to utilize the hearing aids' onboard directional microphones in conjunction with a remote microphone gives listeners the benefits of remote microphone use without sacrificing nearfield intelligibility. The Roger system has also been shown to improve cell phone communication amongst cochlear implant patients.

Despite demonstrated advantages, use of remote microphone assistive devices among adults is low. In a recent study of listeners with severe hearing loss-a group which has substantial difficulty communicating in background noise, and is likely to receive significant benefits from remote-microphone devices-less than 10% reported use of a remote microphone. While cost may be a barrier for some users, even when such systems are available for free (as in the Veterans Administration), use is still low. One reason may be uncertainty among both providers and potential users as to expected benefit for a given listener. For example, Lewis et al. failed to demonstrate a clinically-significant benefit of remote microphone use using a work-life outcomes scale in a cohort of mostly nonworking (retired) participants. Wolfe et al. found significant improvements in objective speech recognition on average, but with a wide range of benefit (from 10% to 60% improvement across individual participants). That study also suggested that individual factors may affect remote microphone benefit, in that the magnitude of improved recognition was correlated with the ability to use spatial cues to improve recognition.

Research Locations:

All study tasks will take place in the Hearing Aid Lab and/or Northwestern's Center for Audiology, Speech, Language and Learning.

When testing in the Hearing Aid Lab, Frances Searle building room 1-451, we will either use the sound booth or lab space. All hearing related tasks take place in a sound booth which is a sound treated 8'x 8' room within the larger lab space. When taking histories or cognitive measures we will use the office space located within the lab or an additional nearby (i.e. same building) testing room. The additional test room is only used if participant confidentiality can be maintained (i.e. conversation is not audible to those outside the room). When using the Center for Audiology, Speech, Language and Learning all tasks will take place in a sound proof booth, in a clinical Hearing Aid fit room, or the virtual sound environment (ViSoR). ViSoR is a 16' by 14' by 9' space capable of simulating the acoustics and background noise properties of any environment by using an array of speakers.

Approach

The trial will use a within-subjects design consisting of baseline assessment (see assessments), hearing aid with Roger connect fitting, a four week trial period of use in the participant's everyday environment(s), and outcome measures.

Participants who qualify for a dome fitting will start their trial the same day as their baseline assessment. Participants who require a custom mold fitting will have earmold impressions taken at their baseline assessment and then be fit with the trial devices after the custom earmold has arrived back in the lab, usually about one week later. During an earmold impression the ear is visually inspected with an otoscope (magnifying scope with light). A cotton block and soft material are placed in the ear. The resulting impression created by the soft material is used to order an earmold for later testing. This is a standard clinical procedure.

A licensed clinical audiologist will perform the assessments, fitting and counseling of hearing aids and Roger system, and conduct the outcome measures. To ensure appropriate fit and use by the participants, there will be a follow-up one week after being fit with the devices. During this appointment participants will be evaluated and their hearing aid logging will be checked for compliance.

Hearing aid/Roger fitting: Trial hearing aids and clinically-appropriate earmolds or domes will be provided by Phonak at no charge to the participants for the duration of the trial. Those aids are expected to be drawn from Phonak's advanced technology level and to provide datalogging via 7 base programs. Aids will be set to NAL-NL2 targets using probe microphone measurements. Directional microphones will be enabled and verified via probe-microphone testing. Roger will be verified via probe-microphone testing, following clinical best practice. Appropriate hearing aid adjustments (as judged by the study audiologist) will be permitted to provide acceptable sound quality and loudness. Final REARs will be recorded. The study audiologist will instruct participants regarding hearing aid and Roger device use. PHAST-R and a Roger competency questionnaire (to be developed with input from Phonak) will be used to document understanding of device function at the fitting and one week follow-up appointments. Participants will then wear the hearing aids and use the Roger system for 1 month in their everyday listening environments. At the completion of the trial, participants will return to the lab for outcome assessments and to provide spontaneous feedback regarding their experiences. Hearing aids and remote microphone will be returned to the study site following completion of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18-85 years
2. Speak English as their primary language
3. Normal or corrected to normal vision
4. Sensorineural hearing loss with pure-tone thresholds 20-85 dB HL at octave frequencies between 500 and 3000 Hz
5. Current hearing aid wearer with at least 3 months of experience

Exclusion Criteria:

1. Clinically significant unstable or progressive medical conditions, or conditions which, in the opinion of the investigator places the participant at unacceptable risk if he or she were to participate in the study
2. Participants who do not pass a cognitive screening test (e.g., MoCA)
3. Significant history of otologic or neurologic disorders
4. Conductive hearing loss pathology or fluctuating hearing loss

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Souza, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experienced Hearing Aid User: Single arm study, all participants in this arm. Participants will be experienced hearing aid users.
  Remote Microphone: Experienced hearing aid users will be trained on and use a remote microphone for 30 days. Pre- and Post- measures will be taken to determine benefit. Participant characteristics will also be assessed (such as self-efficacy) to explore personality factors that may contribute to benefit from devices.
Period: Overall Study
Arm/Group | Experienced Hearing Aid User
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experienced Hearing Aid User
Number analyzed (Participants) | 22
Age, Continuous [Mean (Full Range); unit: years] | 75.5 [59 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Abbreviated Profile of Hearing Aid Benefit (APHAB) [Mean (Full Range); unit: % of problems] — The APHAB is a questionnaire administered before and after intervention asking a lister to rate how much difficulty they have in different listening scenarios. An overall and 4 subscores (Background noise, Ease of Communications, Aversiveness, and Reverberation) are then calculated based on the responses. Population: Participants who did not complete their study participation prior to the start of Covid shutdown are excluded, as their opportunity for social activity and listening environments drastically changed from their baseline measurements.
  % of problems
    APHAB: Overall Baseline: number analyzed (Participants) | 17
    APHAB: Overall Baseline | 28.9 [10.1 to 47.0]
    APHAB Background Noise Baseline | 37.0 [10.5 to 64.3]
    APHAB Aversiveness Baseline | 39.7 [1.0 to 85.00]
    APHAB Ease of Communication Baseline | 20.15 [2.8 to 49.8]
    APHAB Reverberation Baseline | 30.4 [4.7 to 66.5]
% of words repeated correctly in a sentence recog. task with variable levels of background noise: HA [Mean (Standard Deviation); unit: % Correct] — Participants listened to a series of sentences presented in variable background noise. They repeated each sentence to the best of their abilities. They are scored based on the number of key words (5 in each sentence) they get correct. Population: Participants who did not complete their study participation prior to the start of Covid shutdown are excluded, and their opportunity for social activity and listening environments drastically changed from their baseline measurements.
  % Correct
    number analyzed (Participants) | 17
    (all) | 61.0 (35.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: Self assessment, disability based inventory that is used to document outcomes of hearing aid fittings. The APHAB uses a percentile scale (Percent of Problems). This measure has 4 subscales: Ease of communication (EC), Reverberation (RV), Background Noise (BN), and Aversiveness (AV). A lower score indicates a better outcome. We will look at both the global change (defined as EC, RV, and BN scores improving by at least 5 points each) and individual subscales (For EC, RV, or BN a change in 22 points is considered significant and for AV a change of 31 points is needed to be considered significant).
Time Frame: Change from baseline to final appointment will be assessed. Participants will take a baseline at the start of the trial and then complete post-intervention at the end of the 30-day trial.
Population: Participants who did not complete their study participation prior to the start of Covid shutdown are excluded, as their opportunity for social activity and listening environments drastically changed from their baseline measurements.
Measure: Mean (Full Range); unit: % of Problems (Change from baseline)
Arm/Group | Experienced Hearing Aid User
Number analyzed (Participants) | 17
% of Problems (Change from baseline)
  Overall APHAB Change | 7.64 [-11.7 to 24.8]
  Change in BN | 12.5 [-5.8 to 35.1]
  Change in RV | 4.8 [-22.8 to 37.7]
  Change in EC | 6.3 [-1.5 to 23.7]
  Change in AV | -2.6 [-70.3 to 35.2]

2. Secondary Outcome: Change in Speech, Spatial, and Qualities of Hearing (SSQ)
Description: Questionnaire, clinical patient interview design where participants respond on a scale of 0 to 10, with 10 indicating perfect hearing ability and 0 indicating complete inability.There are 3 subscales calculated by averaged the responses to the questions for each subscale. A change of 2 points is considered a moderate effect with increase in score indicating improvement.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Experienced Hearing Aid User
Number analyzed (Participants) | 17
score on a scale
  Speech | 1.7 [0 to 3.6]
  Spatial | 0.6 [-0.9 to 5.1]
  Quality | 1.1 [-1.2 to 4.9]

3. Secondary Outcome: % of Words Repeated Correctly in a Sentence Recognition Task With Variable Levels of Background Noise
Description: Participants had to repeat sentences presented to them in varying levels of background noise. Sentences are scores based on the number of key words (5) they get correct.
Time Frame: End of trial: Objective speech intel was collected in one session at the end of the 30 day trial with the remote microphone. Order of conditions (Hearing aid only and Hearing Aid+ Remote Mic) was randomized.
Population: as for outcome 1
Measure: Mean (Full Range); unit: % Correct
Arm/Group | Experienced Hearing Aid User
Number analyzed (Participants) | 17
% Correct
  Hearing Aid Only | 60.0 [0 to 100]
  Hearing aid + Remote Mic | 82.7 [0 to 100.00]

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Experiences Hearing Aid User
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03897634/Prot_001.pdf